CLINICAL TRIAL: NCT06734169
Title: Depression Among Cardiothoracic Patients in Baghdad: A Cross-Sectional PHQ-9 Study
Brief Title: Depression Among Cardiothoracic Surgery Patients in Baghdad
Acronym: PHQ-9
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241210C; 011 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Depression
Keywords: PHQ-9
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This observational study aims to estimate the prevalence and severity of depression among patients in the Cardiothoracic Surgery Ward in Baghdad City, Iraq, using a self-administered PHQ-9 questionnaire. The main questions it aims to answer are:

What is the prevalence of depression among cardiothoracic surgery patients? How is the severity of depression distributed within this group? Are there specific environmental or demographic factors associated with higher levels of depression?

Participants will:

Fill out the PHQ-9 in order to measure the severity of depressive symptoms at a specific moment in time.

Demographic and clinical variables such as age, gender, socioeconomic status, surgery type, comorbidities, and hospital stay length should be taken to look for a possible relationship with depression.

DETAILED DESCRIPTION:
Depression is a common mental health condition that frequently coexists with chronic illnesses and surgical conditions, including cardiothoracic surgeries, significantly impacting recovery and long-term health outcomes. Studies have established a link between depressive symptoms and adverse postoperative results, including prolonged hospital stays, decreased quality of life, and increased mortality rates. In surgical populations, depression often remains undetected and untreated, exacerbating its negative effects on patient outcomes.

In Iraq, particularly in Baghdad, the prevalence of depression among cardiothoracic surgery patients is not well documented. The region's ongoing socio-economic challenges, coupled with limited access to mental health resources, pose additional barriers to adequate psychological care. Addressing these challenges requires robust data to inform targeted interventions.

The Patient Health Questionnaire-9 (PHQ-9) is a validated and widely used tool for screening depression in clinical and nonclinical populations It consists of nine questions that assess the frequency of depressive symptoms over the past two weeks, with scores ranging from 0 to 27. Diagnostic Cut-off: A score of ≥10 is often used as a threshold for identifying major depressive disorder with a high degree of sensitivity and specificity. Additionally, changes in PHQ-9 scores over time are used to evaluate the effectiveness of treatment. Its applicability in diverse populations makes it suitable for assessing depression among cardiothoracic surgery patients in Baghdad .

Baghdad is a region with limited local data on mental health, making it crucial to understand the mental health burden in surgical populations. This study aims to investigate the prevalence and severity of depression in this patient group, providing critical insights to bridge the gap in mental health care and improve surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the cardiothoracic surgery ward.
* Patients who are able to understand and provide informed consent.
* Patients who have the cognitive ability to complete the PHQ-9 questionnaire.

Exclusion Criteria:

* Patients with a history of diagnosed psychiatric disorders other than depression.
* Patients who are critically ill or in a life-threatening condition and unable to participate.
* Patients who are unable to understand the PHQ-9 questionnaire due to language or cognitive barriers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (18 years and older) admitted to the cardiothoracic surgery ward at Al-Kadhimiya Teaching Hospital in Baghdad.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Depression | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  Proportion of cardiothoracic surgery patients at Al-Kadhimiya Teaching Hospital who exhibit depressive symptoms.
Severity of Depression | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The severity of depression in this study will be determined based on the scores obtained from the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 categorizes depression severity as follows:
  Minimal depression: Scores 0-4, indicating little to no symptoms. Mild depression: Scores 5-9, suggesting occasional symptoms that may not significantly affect daily functioning.
  Moderate depression: Scores 10-14, indicating more frequent symptoms that can interfere with daily life.
  Moderately severe depression: Scores 15-19, showing pronounced symptoms that significantly impact daily activities.
  Severe depression: Scores 20-27, with symptoms that are debilitating.
Patient Health Questionnaire-9 (PHQ-9) | Data collection will occur over a 3-months period, with each participant completing the PHQ-9 assessment at a single point during this time frame.
  The total score can range from 0 to 27. Higher scores indicate greater severity of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCormick KM, Naimark BJ, Tate RB. Uncertainty, symptom distress, anxiety, and functional status in patients awaiting coronary artery bypass surgery. Heart Lung. 2006 Jan-Feb;35(1):34-45. doi: 10.1016/j.hrtlng.2005.08.002. PMID 16426934
- [Background] Underwood MJ, Firmin RK, Jehu D. Aspects of psychological and social morbidity in patients awaiting coronary artery bypass grafting. Br Heart J. 1993 May;69(5):382-4. doi: 10.1136/hrt.69.5.382. PMID 8518057
- [Background] Tully PJ, Baker RA. Depression, anxiety, and cardiac morbidity outcomes after coronary artery bypass surgery: a contemporary and practical review. J Geriatr Cardiol. 2012 Jun;9(2):197-208. doi: 10.3724/SP.J.1263.2011.12221. PMID 22916068
- [Background] Morys JM, Bellwon J, Hofer S, Rynkiewicz A, Gruchala M. Quality of life in patients with coronary heart disease after myocardial infarction and with ischemic heart failure. Arch Med Sci. 2016 Apr 1;12(2):326-33. doi: 10.5114/aoms.2014.47881. Epub 2015 Jan 14. PMID 27186176
- [Background] Tully PJ, Baker RA, Winefield HR, Turnbull DA. Depression, anxiety disorders and Type D personality as risk factors for delirium after cardiac surgery. Aust N Z J Psychiatry. 2010 Nov;44(11):1005-11. doi: 10.3109/00048674.2010.495053. PMID 21034183
- [Result] Stenman M, Sartipy U. Depression Screening in Cardiac Surgery Patients. Heart Lung Circ. 2019 Jun;28(6):953-958. doi: 10.1016/j.hlc.2018.04.298. Epub 2018 May 16. PMID 29871802
- [Result] Manea L, Gilbody S, McMillan D. Optimal cut-off score for diagnosing depression with the Patient Health Questionnaire (PHQ-9): a meta-analysis. CMAJ. 2012 Feb 21;184(3):E191-6. doi: 10.1503/cmaj.110829. Epub 2011 Dec 19. PMID 22184363
- [Result] Sadik S, Bradley M, Al-Hasoon S, Jenkins R. Public perception of mental health in Iraq. Int J Ment Health Syst. 2010 Oct 11;4:26. doi: 10.1186/1752-4458-4-26. PMID 20937100
- [Result] Murphy BM, Elliott PC, Higgins RO, Le Grande MR, Worcester MU, Goble AJ, Tatoulis J. Anxiety and depression after coronary artery bypass graft surgery: most get better, some get worse. Eur J Cardiovasc Prev Rehabil. 2008 Aug;15(4):434-40. doi: 10.1097/HJR.0b013e3282fbc945. PMID 18677168
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941